CLINICAL TRIAL: NCT07195461
Title: A Feasibility Study Evaluating the Magnetic Bead Tracking System and Its Safety and Effectiveness When Used With a Bionic External Prosthesis to Improve Prosthetic Controllability for Persons With Transtibial Amputation
Brief Title: Feasibility Study Evaluating the Safety and Effectiveness of Magnetic Bead Tracking System When Used With a Bionic External Prosthesis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: MuscleMetrix, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001485
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Transtibial Amputee; Transtibial Amputation
Keywords: transtibial; amputation; amputee; magnet; prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transtibial amputees (Experimental): Up to five subjects signing an informed consent and meeting all inclusion and exclusion criteria will be enrolled into the study to receive the Magnetic Bead Tracking System. Each subject will serve as their own control in a repeated measures ('within subjects') design. During experimentation, each subject will have prosthetic gait performance measured while using the Magnetic Bead Tracking System compared to an intrinsic robotic controller.
  Interventions: Device: Magnetic Bead Tracking System

INTERVENTIONS:
Device: Magnetic Bead Tracking System — The Magnetic Beads will be implanted in a subject during either an already required revision of an existing unilateral or bilateral transtibial amputation or during the performance of a unilateral or bilateral transtibial amputation.

SUMMARY:
The investigation is an early feasibility study in up to 5 subjects, in which the primary objective is to capture preliminary safety and effectiveness information on the Magnetic Bead Tracking system.

DETAILED DESCRIPTION:
This is an early feasibility study designed to provide preliminary evidence for the safety and effectiveness of the Magnetic Bead Tracking System for the control of a one degree-of-freedom (DoF) ankle-foot prosthesis at the transtibial amputation level on up to N=5 study subjects. Each subject will serve as their own control in a repeated measures ('within subjects') design. During experimentation, each subject will have prosthetic gait performance measured while using the Magnetic Bead Tracking System compared to an intrinsic robotic controller.

The Magnetic Bead Tracking System consists of pairs of magnetic beads, and a set of magnetic field sensors that are intended to measure and track the length of muscles and the speed at which they move in real-time. The system uses multiple pairs of implanted magnetic beads to track tissue strains via an array of externally worn magnetic field sensors, which senses the relative locations of the implanted magnetic beads. When implanted in muscle in the residual limb of an amputee, the muscle length signal is used as an indicator of human intent and is conveyed to a robotic prosthesis, providing heightened, natural, reflexive control of prosthetic limbs in subjects with transtibial amputation. Specifically, in the proposed study, the system will be used with a computer controlled, powered ankle prosthesis to provide sensory position, speed, and force data to increase the accuracy of neuromuscular control models and allow for intuitive, simultaneous position and torque control of the prosthesis.

Safety of the Magnetic Bead Tracking System will be evaluated throughout the study by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device. Adverse events with clinical signs or symptoms will be collected when volunteered by subjects and/or observed by Investigators. Serious Adverse Events will be reported on a per event and per subject basis up to 6 months. At each study visit, the subject will be asked to report any issues, and will have a comprehensive examination of the affected limb performed by study physicians and/or trained staff.

Due to the small number of subjects, this study will be treated as a case study. For each case, information, such as demographic and subject information, adherence to the study protocol, safety, and performance data will be collected and described. At the end of the study, each case will be evaluated, and a determination will be made, as to whether (1) any unanticipated adverse device effects and/or revisions/removals of the device occurred, and (2) the study objective was met for that particular case.

For each case, variables will be summarized qualitatively by visit and (where applicable) by difference from pre-op assessment and post-op assessments. This assessment will be performed separately for each case. In addition, a quantitative measurement of preferred walking speed will serve as a primary variable for the evaluation of system performance in AIM 1, and the time to traverse an obstacle course will serve as a primary variable for AIM 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 22-65 at the time of surgery.
* The patient must already have an existing unilateral or bilateral transtibial amputation requiring revision or a medical condition requiring performance of a unilateral or bilateral transtibial amputation.
* If the patient does not already have an amputation, the patient must have undergone independent consultation with a lower extremity surgical specialist to ensure they have exhausted all limb salvage options prior to undergoing amputation, as well as a psychiatric evaluation to ensure appropriate capacity and volition, and a pain medicine evaluation to ensure that all pain control options outside of amputation have been addressed.
* The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above, as determined by a trained and certified prosthetist and confirmed by study investigators, through use of a patient history and physical examination).
* The patient must have adequate soft tissue bulk and muscle mass present in the operative limb to support appropriate wound healing.
* The patient must demonstrate volitional activation of the muscles into which magnet placement is intended.
* In the opinion of the investigator, the patient must likely be able to tolerate the pressure of a prosthetic socket during ambulation post-operatively.
* In the opinion of the investigator, the patient must have absence of any physical limitations, addictive diseases or underlying medical conditions that may preclude the patient from being a good study candidate.
* The patient must have willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.
* The patient must have willingness and ability to provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with any active skin disease in the subject limb.
* Patients with severe comorbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the patients to be a good study candidate (i.e., other disease processes, mental capacity, substance abuse, shortened life. expectancy, vulnerable patient population, etc.).
* Patients with the following concurrent diseases: active infection or dormant bacteria, metabolic bone disease and/or metastatic lesions in the residual tibia.
* Patients weighing over 285 lbs. with the prosthesis, at time of screening.
* Patients for whom skeletal growth is not complete. Completed skeletal growth is defined through the finding of generally closed epiphyseal zones on X-ray.
* Patients with advanced atrophic muscle and/or compromised soft tissue coverage in the operative limb.
* Patients with evidence of or a documented history of severe peripheral vascular disease, diabetes mellitus (type I or type II), skin diseases, neuropathy or neuropathic disease and severe phantom pain, or osteoporosis, such that, in the opinion of the investigator, will not allow the patient to be a good study candidate.
* Patient with a history of systemically administered corticosteroids, immune-suppressive therapy or chemotherapy drugs within six (6) months of implant surgery.
* Patients with a known need of future MRIs.
* Patients currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study.
* Active smokers will be excluded from candidacy; those patients willing to undergo tobacco cessation will need to be completely abstinent from tobacco use for at least 6 weeks preoperatively.
* Women who are pregnant, lactating or planning a pregnancy during the first twelve (12) months of the post-surgical follow-up.
* Patient having an allergy to any component of the device.
* Patients with concurrent illness, disability or geographical residence that would hamper attendance at required study visits.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Walking Speed | One timepoint, between days 150-180.
  The preferred and fastest walking speeds across level-ground and uneven walking surfaces will be measured as the primary study variables for AIM 1. To make these measurements, the time duration will be measured for each study subject to walk at steady state speed overground across 10m walkways at their preferred and fastest walking speeds. Subjects will receive standardized instructions encouraging them to either walk at their comfortable walking speed, or at their maximum walking speed, across each level-ground andan uneven 10m walkway. The investigators expect that the preferred and maximum speeds will be higher when employing the magnetomicrometry (MM) prosthetic controller compared to the commercial intrinsic controller, in support of the H1 hypothesis.
Obstacle course speed | One timepoint, between days 150-180.
  The time to traverse an obstacle course will be evaluated to test obstacle avoidance, changes in walking direction, slope/stair variations, and speed transients, testing the ability of each controller to deliver rapid gait maneuvers while subjects walk across the unstructured environment. The investigators expect that the time to complete the obstacle course will be lower when employing the MM controller compared to the commercial intrinsic controller, further supporting the H1 hypothesis.

SECONDARY OUTCOMES:
Walking Distance | One timepoint, between days 150-180.
  The Six Minute Walk Test (6MWT) across a level-ground surface will be evaluated, or the maximum distance a person can walk in a six-minute period. Using an indoor track, the total distance each subject can walk throughout a six-minute interval will be measured for each controller (magnetomicrometry (MM) vs. Intrinsic). The investigators expect that the 6MWT will be higher when employing the MM prosthetic controller compared to the commercial intrinsic controller, further supporting the H1 hypothesis.
Gait Symmetry | One timepoint, between days 150-180.
  Asymmetry between the double-support time preceding intact limb (tdspi) and preceding prosthetic limb (tdsip) transitions will be measured on level ground and slopes (instrumented treadmill), and for stair ascent and descent. The investigators expect that a composite measure of Gait Symmetry will demonstrate the best performance when the powered ankle-foot prosthesis is controlled using the MM controller, further supporting the H1 hypothesis.
Biologic Realism | One timepoint, between days 150-180.
  Prosthetic and unaffected leg ankle net-work, wA , will be measured as defined in [2] on level ground and slopes (instrumented treadmill), and for stair ascent and descent. The investigators expect that the net-work measures when employing the MM controller will more closely match that of the contralateral intact ankle than compared to the commercial intrinsic controller, further confirming the H1 hypothesis.
Musculoskeletal Stress | One timepoint, between days 150-180.
  Bilateral knee moments will be measured as defined in on level ground and slopes (instrumented treadmill). The investigators expect the contralateral knee adduction moment measure of musculoskeletal stress to be lowered when employing the MM controller as compared with the intrinsic controller, further supporting the H1 hypothesis.
Stability (1) | One timepoint, between days 150-180.
  Posturographic parameters will be derived from pelvic center of mass (COM) position collected as subjects stand on a one axis (anteroposterior) balance board. The investigators expect that stability metrics will show the best performance when the powered ankle-foot prosthesis is controlled using the MM interface as compared with the intrinsic controller, further supporting the H1 hypothesis.
Relative pain levels | One timepoint, between days 150-180.
  The relative pain levels experienced by the user at the unaffected knee and lower back will be assessed using a Visual Analogue Scale (VAS, 0 to 10). The investigators expect a lower pain score when the powered ankle-foot prosthesis is configured for the MM controller as compared with the intrinsic controller, further supporting the H1 hypothesis.
General Mobility | One timepoint, between days 150-180.
  Patient-reported mobility will be assessed as measured by the Prosthetic Limb Users Survey of Mobility (PLUS-M). The investigators expect a score of greater than or equal to 5 when using the MM controller, indicating a significant improvement in mobility compared to the commercial intrinsic controller.
Embodiment | One timepoint, between days 150-180.
  Patient-reported embodiment will be assessed as measures by the Prosthesis Embodiment Scale for Lower Limb Amputees (PEmbS-LLA). PEmbS-LLA is a 10-item, patient-reported questionnaire (using a 7-point Likert scale) designed to measure how well a lower limb amputee integrates their prosthesis into their body representation and sense of self.The investigators expect a higher level of embodiment when using the MM controller compared to the commercial intrinsic controller.
Stability (2) | One timepoint, between days 150-180.
  Equilibrium scores, limits of stability, symmetry, and latency and amplitude of response to perturbation will be assessed from Computerized Dynamic Posturography (CDP). The investigators expect that stability metrics will show the best performance when the powered ankle-foot prosthesis is controlled using the MM interface as compared with the intrinsic controller, further supporting the H1 hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Carty, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.